CLINICAL TRIAL: NCT04711096
Title: Ultrasound-guided Transversus Abdominis Plane (TAP) Block Versus Local Wound Infiltration for Post-operative Analgesia After Cesarean Section Under General Anesthesia.
Brief Title: Ultrasound-guided TAP Block Vs Local Wound Infiltration for Analgesia After Cesarean Section.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mostafa R Bakry, Master's Degree, The principal investigator, Ain Shams Maternity Hospital
Other Study IDs: Post Cesarean TAP Block
Record Dates: First submitted 2021-01-08; First posted 2021-01-15 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain Control
Keywords: Post Cesarean TAP Block; TAB block; Postoperative Pain control
MeSH Terms: interventions — Dental Occlusion; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: TAB group formed of 65 patients
  Interventions: Procedure: Ultrasound-guided transversus abdominis plane (TAP) block 0.25% bupivacaine.
- Group B: Group B : The Infiltration Group formed of 65 patients.
  • This group will B wills provided with single-shot local anesthetic wound infiltration with 20 ml of 0.25% bupivacaine injected subcutaneously above and below skin incision before closure of skin.
  Interventions: Procedure: Ultrasound-guided transversus abdominis plane (TAP) block 0.25% bupivacaine.
- Group C: Group C : Narcotics only group formed of 20 patients
  • routine analgesic was taken only without any intervention

INTERVENTIONS:
Procedure: Ultrasound-guided transversus abdominis plane (TAP) block 0.25% bupivacaine. — After preparing the skin with antiseptic solution, a linear high frequency ultrasound probe will be placed abdominal wall between the iliac crest and the costal margin. A Spinal needle 22g attached with flexible tubing to a syringe filled with saline will be used to perform the block then introduced through the skin anteriorly in the plane between the internal oblique and transversus abdominis muscles with its tip lying in the mid axillary line. To assist with identifying these structures, The final position of the probe will to be no further anterior than the anterior axillary line. If satisfactory views are not obtained, the TAP block will not be performed. Hydro dissection with saline (2-5 ml) will be used to separate the fascial layers. After aspiration to exclude inadvertent vascular puncture, 20 ml of the 0.25% bupivacaine will be injected . TAP block will be performed in a similar fashion on the opposite side.
  Other Names: local wound infiltration
  Groups: Group A; Group B

SUMMARY:
Adequate pain control after cesarean delivery is a major concern for both parturients and obstetrician, and it usually comprise a combination of systemic and regional techniques. The transversus abdominis plane (TAP) block, affecting the nerves supplying the anterior abdominal wall, is a recently introduced, promising regional analgesic technique for a variety of abdominal and pelvic surgeries including cesarean delivery .

Infiltration of local anesthetic into the surgical wound (either as a single shot or using indwelling catheters) has long been used for postoperative analgesia, Both the TAP block and wound infiltration, are superior to placebo, however, it is unknown which of them provides better analgesia after cesarean delivery because of a scarcity of randomized clinical trials.

This study aimed to compare bilateral US guidedTAP block with single-shot local anesthetic wound infiltration for analgesia after cesarean delivery performed under general anesthesia. The investigators hypothesized that the TAP block would decrease postoperative cumulative opioid consumption at 24 hours.

DETAILED DESCRIPTION:
The Anaesthesilogist is Senior staff trained on such procedure.

* Pre-operative settings
* The study subjects will randomly assigned to 3 equal groups (TAP group, infiltration group and narcotics only group ) using a computer-generated table of random numbers. A single investigator will assess the patients for eligibility, obtained written informed consent, and record the baseline data for each participant before delivery. Sequentially numbered, sealed opaque envelopes containing group allocation will be opened by the primary investigator after administration of general anesthesia . Neither the study subjects nor the outcome assessors knew the study group
* Routine preoperative investigations will be done to all patients including laboratory investigations as (complete blood picture, liver function tests, prothrombin time and partial thromboplastin time).
* Demographic data as age, weight, will be recorded.

All mothers who scheduled for elective cesarean delivery who fulfilled inclusion criteria and volunteer are assessed by:

Postoperative pain by Numerical Rating Scale (NRS) pain score (range, 0-10; 0, no pain; 10, worst pain) on arrival in the post-labor ward (time 0) and at 2,4,6, 8, 12,18 and 24 hours postoperatively.

The duration of block (defined as the interval between performing the block and the time of the first request for analgesia) and total pethidine consumption were recorded in the 24 hours after surgery The level of patient satisfaction was measured numerically by a Likert scale ranging from one to five, 1: "not satisfied at all," 2: "slightly satisfied," 3: "moderately satisfied," 4: "very satisfied," and 5: "highly satisfied". Any adverse effects or complications will be recorded.

* Wide bore venous access will be secured by 18 G intravenous canula
* The procedure is done in the operating rooms (OR) under complete aseptic technique with prophylactic antibiotics (e.g. 2 gm ceftriaxone).

Intra-operative Setting

* The patient will be monitored during the procedure using pulse oximetry, non-invasive blood pressure & ECG and capnography
* Patients receive General anesthesia induction by propofol (2mg/kg),Rocuronium(0.5mg /kg) for rapid sequence intubation& Fentanyl (1 mcg /kg)
* Maintenance with rocuronium & isoflurane 1.2%
* Equipment's that will be used for each patient are:
* Sterile towels, sponges, 4-inch gauze packs and povidone iodine 10% for sterilization
* Sterile gloves, marking pen, 18-gauge cannula and 10-ml syringes containing drugs for administration of the procedure.Ultrasound device with Linear probe with high frequency (6 -13 MHz) will be used in imaging of patient
* drugs that will be used In our study are: A 20 ml vial of 0.5% Bupivacaine HCl , pethidine IV (50-150 mg)
* Lower segment cesarean section will be performed using the Pfannenstiel incision
* An anesthesiology resident will administer the general anesthesia, will record the intraoperative data (the duration of surgery), and prepared, as instructed by the primary investigator , the local anesthetic solution for the TAP block and wound infiltration. The outcome data (pethidine consumption, time to the first pethidine dose, pain scores level , side effects, and patient satisfaction) will be recorded by a blind investigator who will visite the patient in the ward at 2, 4, 6, 12, and 24 hours postoperatively.

Group A: TAB group formed of 65 patients

* After completion of LSCS and skin closure and while the patient is still on the operating table U/S guided TAP block will be done using the following procedure:
* After preparing the skin with antiseptic solution, a linear high frequency ultrasound probe (Superficial probe of mindray DP-20) will be placed transversely on the anterolateral abdominal wall between the iliac crest and the costal margin. Under US guidance, the three layers of muscles -external oblique, the internal oblique, and the transversus abdominis will be identified. A Spinal needle 22g attached with flexible tubing to a syringe filled with saline will be used to perform the block. The needle will be then introduced through the skin anteriorly in the plane of the ultrasound beam and advanced into the fascial plane between the internal oblique and transversus abdominis muscles with its tip lying in the mid axillary line. To assist with identifying these structures, the probe will be moved anteriorly to the rectus sheath and the fascial planes followed laterally. The final position of the probe will to be no further anterior than the anterior axillary line. If satisfactory views are not obtained, the TAP block will not be performed. Hydro dissection with saline (2-5 ml) will be used to separate the fascial layers. After aspiration to exclude inadvertent vascular puncture, a test dose of 1-2 ml of the drug will be injected to confirm needle placement. After a negative test dose, 20 ml of the 0.25% bupivacaine will be injected while closely observing for signs of toxicity e.g CVS toxicity which may be in form of early features e.g hypertension, tachycardia and ventricular arrhythmia or may be in form of late features e.g hypotension, bradycardia, heart block and decreased contractility and other toxic signs e.g tinnitus, perioral numbness, metallic taste in mouth, slurring of speech and mental status changes). TAP block will be performed in a similar fashion on the opposite side.

Group B : The Infiltration Group formed of 65 patients.

• This group will B wills provided with single-shot local anesthetic wound infiltration with 20 ml of 0.25% bupivacaine injected subcutaneously above and below skin incision before closure of skin.

Group C : Narcotics only group formed of 20 patients • routine analgesic was taken only without any intervention

Post operative settings:

* At the end of the surgery and complete recovery from anesthesia, the patient will be kept under observation postoperatively for 4 hours to monitor vital signs (conscious level, blood pressure, heart rate, respiratory rate and pattern & any possible limb weakness or abnormal sensation) then discharged to ward & observed to be followed for returning of pain.
* Duration of surgery (time from the start of skin incision to the end of skin closure) will be recorded. All the study subjects will receive postoperative standard analgesia (30 mg of IV ketorolac every 8 hours starting immediately after surgery and 1 gm of oral paracetamol every 6 hours starting 4 hours after surgery with caution to toxic dose) .
* The patients will be observed for the occurrence of any adverse effect and/or complication related to the procedure (e.g. hematoma), or to the study drugs (e.g. hypotension/hypertension (i.e. 20% decrease or increase from the baseline value), bradycardia (HR <50 beats/min) or tachycardia (HR > 120 beats/min), nausea, vomiting, and hypoxemia (SpO2 <90%)).
* Assessment of pain involves asking a patient to rate her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 equal to the worst possible pain after first hour, 2nd hour,4th hour, 6th hour, 12th hour and 24th hour at wards after end of surgery.

Pain is usually managed by pethidine IV based on patient complain. the analgesic dose of pethidine will be 50 mg to be repeated on demand (NRS >4) provided that the total 24 hour dosage will not exceed 150 mg . At recovery room mothers asked to report their pain based on 11 point NRS score during first 24 hour. Patient satisfaction from postoperative analgesia will be assessed at 24 hours postoperatively using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied,and 5 = very satisfied) after first hour, 2nd hour,4th hour, 6th hour, 12th hour and 24th hour at wards after end of surgery.

• A time in minutes from end of surgery to first analgesia request were documented together with total analgesia consumed in the first 24 h. In addition, incidence of postoperative nausea and vomiting will be documented within 24 h.

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing elective cesarean section under general anathesia

  * Pfannenstiel Skin Incision
  * Age between 18 and 40 years old
  * BMI between 18 and 35 kg/m2

Exclusion Criteria:

* • Patient refusal.

  * BMI<18 kg/m2 or>35 (require different dose of analgesia)
  * Height <150 or > 180 cm (require different dose of analgesia)
  * Patients with any neurological deficit due to neuropathy and pain score affection
  * Patients with bleeding disorders which may lead to hematoma
  * HTN (Vasculopathy which can lead to hematoma).
  * Cardiac disease ( Vasculopathy on anticoagulant which can lead to hematoma)
  * DM (decrease systemic and local immunity which can lead to abscess at injection site and due to neuropathy and pain score affection).
  * Liver disease (defective clotting factors).
  * A history of relevant drug allergy or Hypersensitivity to any of the drugs used in the study due to impair of proper follow up of pain postoperative
  * History of recent opioid exposure due to affection on pain score
  * Local skin infection due to abscess formation
  * Obstetric complications e.g placenta previa and rupture uterus due to extensive tissue damage and dissection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study subjects will randomly assigned to 3 equal groups (TAP group and infiltration group and Narcotics only group) of patients undergoing elective cesarean section under general anathesia in Ain Shams Maternity hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain severity assessed by the Numerical Rating Scale (NRS) pain score at 1,2,4,6, 12, and 24 hours | 24 hours after the procedure
  Assessment of pain involves asking a patient to rate her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 equal to the worst possible pain after first hour, 2nd hour,4th hour, 6th hour, 12th hour and 24th hour at wards after end of surgery.
The duration of analgesia achieved by each type of block assessed by the time of first postoperative pethidine dose required. | 24 hours after the procedure
  By asking the patients about the first time to analgesic request

SECONDARY OUTCOMES:
Cumulative pethidine consumption at 2, 4, 6, and 12 hours, NRS at 0, 4, 6, 12, and 24 hours. | 24 hours after the procedure
  By observation of first time to analgesia requested.
the incidence of side effects and Toxicity (nausea and vomiting and pruritis). | 24 hours after the procedure
  Observation of vital data in the first 24 hours postoperatively.
Patient Satisfaction | 24 hours after the procedure
  Patient satisfaction from postoperative analgesia will be assessed at 24 hours postoperatively using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied,and 5 = very satisfied) after first hour, 2nd hour,4th hour, 6th hour, 12th hour and 24th hour at wards after end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Abdel Rahman, Prof, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adesope O, Ituk U, Habib AS. Local anaesthetic wound infiltration for postcaesarean section analgesia: A systematic review and meta-analysis. Eur J Anaesthesiol. 2016 Oct;33(10):731-42. doi: 10.1097/EJA.0000000000000462. PMID 27259092
- [Result] Bamigboye AA, Hofmeyr GJ. Local anaesthetic wound infiltration and abdominal nerves block during caesarean section for postoperative pain relief. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006954. doi: 10.1002/14651858.CD006954.pub2. PMID 19588413
- [Result] Fusco P, Scimia P, Paladini G, Fiorenzi M, Petrucci E, Pozone T, Vacca F, Behr A, Micaglio M, Danelli G, Cofini V, Necozione S, Carta G, Petrini F, Marinangeli F. Transversus abdominis plane block for analgesia after Cesarean delivery. A systematic review. Minerva Anestesiol. 2015 Feb;81(2):195-204. Epub 2014 Apr 16. PMID 24739207
- [Result] Elamin G, Waters PS, Hamid H, O'Keeffe HM, Waldron RM, Duggan M, Khan W, Barry MK, Khan IZ. Efficacy of a Laparoscopically Delivered Transversus Abdominis Plane Block Technique during Elective Laparoscopic Cholecystectomy: A Prospective, Double-Blind Randomized Trial. J Am Coll Surg. 2015 Aug;221(2):335-44. doi: 10.1016/j.jamcollsurg.2015.03.030. Epub 2015 Mar 27. PMID 25899736
- [Result] Lapmahapaisan S, Tantemsapya N, Aroonpruksakul N, Maisat W, Suraseranivongse S. Efficacy of surgical transversus abdominis plane block for postoperative pain relief following abdominal surgery in pediatric patients. Paediatr Anaesth. 2015 Jun;25(6):614-20. doi: 10.1111/pan.12607. Epub 2015 Jan 9. PMID 25571981
- [Result] Kiran LV, Sivashanmugam T, Kumar VRH, Krishnaveni N, Parthasarathy S. Relative Efficacy of Ultrasound-guided Ilioinguinal-iliohypogastric Nerve Block versus Transverse Abdominis Plane Block for Postoperative Analgesia following Lower Segment Cesarean Section: A Prospective, Randomized Observer-blinded Trial. Anesth Essays Res. 2017 Jul-Sep;11(3):713-717. doi: 10.4103/0259-1162.206855. PMID 28928576
- [Result] Mankikar MG, Sardesai SP, Ghodki PS. Ultrasound-guided transversus abdominis plane block for post-operative analgesia in patients undergoing caesarean section. Indian J Anaesth. 2016 Apr;60(4):253-7. doi: 10.4103/0019-5049.179451. PMID 27141108
- [Result] McDonnell NJ, Keating ML, Muchatuta NA, Pavy TJ, Paech MJ. Analgesia after caesarean delivery. Anaesth Intensive Care. 2009 Jul;37(4):539-51. doi: 10.1177/0310057X0903700418. PMID 19681409
- [Result] Mishriky BM, George RB, Habib AS. Transversus abdominis plane block for analgesia after Cesarean delivery: a systematic review and meta-analysis. Can J Anaesth. 2012 Aug;59(8):766-78. doi: 10.1007/s12630-012-9729-1. Epub 2012 May 24. PMID 22622954
- [Result] Aydogmus M, Sinikoglu S, Naki M, Ocak N, Sanli N, Alagol A. Comparison of analgesic efficiency between wound site infiltration and ultra-sound-guided transversus abdominis plane block after cesarean delivery under spinal anaesthesia. Hippokratia. 2014 Jan;18(1):28-31. PMID 25125948
- [Result] Mudgalkar N, Bele SD, Valsangkar S, Bodhare TN, Gorre M. Utility of numerical and visual analog scales for evaluating the post-operative pain in rural patients. Indian J Anaesth. 2012 Nov;56(6):553-7. doi: 10.4103/0019-5049.104573. PMID 23325940
- [Result] Sharkey A, Finnerty O, McDonnell JG. Role of transversus abdominis plane block after caesarean delivery. Curr Opin Anaesthesiol. 2013 Jun;26(3):268-72. doi: 10.1097/ACO.0b013e328360fa16. PMID 23587731